CLINICAL TRIAL: NCT03310606
Title: Serum and Peritoneal Concentration in Antibiotics During the Surgical Management of Peritonitis: SPAC
Brief Title: Serum and Peritoneal Concentration in Antibiotics During the Surgical Management of Peritonitis
Acronym: SPAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-A00710-53
Record Dates: First submitted 2017-08-28; First posted 2017-10-16 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Peritonitis; Critical Illness
Keywords: Therapeutic drug monitoring
MeSH Terms: conditions — Peritonitis; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peritonitis (Other): Patient received for antibiotic treatment a B lactam according to French recommendation :
  * type of antibiotic : cefotaxime or ceftriaxone or piperacilline/tazobactam or imipenem
  * dose : cefotaxime 2g / cetriaxone 2g / piperacilline 4g / imipenem 1g
  Interventions: Other: Dosage of serum and peritoneal of the B lactam used for antibiotic treatment

INTERVENTIONS:
Other: Dosage of serum and peritoneal of the B lactam used for antibiotic treatment — Dosage of serum and peritoneal of the B lactam used B lactam concerning are : CEFTRIAXONE, CEFOTAXIME, PIPERACILLINE/TAZOBACTAM, IMIPENEM

SUMMARY:
SPAC is a pilote monocentric prospective study about peritonitis and antibiotics pharmacokinetic and pharmacodynamic. The investigators will included 50 patients during 2 years in the University Hospital of Nancy.

The aim of this study is to determine if the beta-lactam dosages recommended by the guidelines for management of intra-abdominal infections (published by the Société française d'anesthésie et de réanimation (Sfar) in december 2015) permitted the achievement of adequatly serum and peritoneal concentrations in the medical and surgical management of peritonitis.

The investigators will collected 3 pairs of serum and peritoneal fluid samples at 3 different times: peritoneal incision, arrival in ICU and 24 hours after admission in ICU in order to compare the concentrations and the minimal inhibitor concentration of bacteria.

The hypothesis is that of a serum and peritoneal antibiotic under dosage.

ELIGIBILITY:
Inclusion Criteria:

* Minimun age limits 18 years
* All sex
* Patients with peritonitis (community or nosocomial) regardless of pathology involved
* Patients treated in the Universty Hospital of Vandoeuvre les Nancy (abdominal surgery unit and surgical Intensive care unit JM Picard)

Exclusion Criteria:

* Beta lactam allergy
* Pregnancy
* Age less than 18 years
* No respect of recommandations for antibiotics ( molecule and dosage)
* Person under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-10-24 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Serum and peritoneal beta lactams concentrations at 3 times | 3 times : Peritoneal incision, Admission in ICU and 24 hours after admission in ICU
  Population : patients with surgical peritonitis. The concentrations are compared with the minimum inhibitory concentrations of bacteria to diagnose a sub therapeutic dosage.

SECONDARY OUTCOMES:
Factors associated with an antibiotic under-dosage | Statistical analysis after 2 years of inclusion
  effect of presence of septic shock on antibiotic concentration
Factors associated with an antibiotic under-dosage | Statistical analysis after 2 years of inclusion
  effect of volume ressucitation on antibiotic concentration
Factors associated with an antibiotic under-dosage | Statistical analysis after 2 years of inclusion
  effect of renal function on antibiotic concentration
Evaluate the relationship between serum and peritoneal concentrations of beta-lactam | Statistical analysis after 2 years of inclusion
  Determination of the antibiotic diffusion coefficient through the peritoneal membrane : difference between serum concentration and peritoneal concentration of B lactam
Morbidity of included patients | Reception on the 8th postoperative day
  Morbidity is assessed by the presence or absence of second peritonitis surgery during hospitalization in ICU and at most 8 days (the mean of the peritonitis stays in the ICU of the investigators in 2016 is 8 days)
Mortality of included patients | Reception on the 8th postoperative day
  The mortality is evaluated by the presence or absence of the death of the patient during the hospitalization in ICU and at most 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel NOVY, MD, Principal Investigator — CHRU NANCY
Locations (1):
- Central Hospital, Vandœuvre-lès-Nancy, France

REFERENCES:
- [Derived] Leon L, Guerci P, Pape E, Thilly N, Luc A, Germain A, Butin-Druoton AL, Losser MR, Birckener J, Scala-Bertola J, Novy E. Serum and peritoneal exudate concentrations after high doses of beta-lactams in critically ill patients with severe intra-abdominal infections: an observational prospective study. J Antimicrob Chemother. 2020 Jan 1;75(1):156-161. doi: 10.1093/jac/dkz407. PMID 31599951